CLINICAL TRIAL: NCT02647034
Title: Using the Stress Ventricular Function Assessment to Evaluate the Long-term Prognosis and Treatment Outcome in Patients With Pulmonary Hypertension
Brief Title: Stress Ventricular Function in Evaluating Patients With Pulmonary Hypertension
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: National Taiwan University Hospital (Other)
Responsible Party: Sponsor
Other Study IDs: 200905040R
Record Dates: First submitted 2015-12-29; First posted 2016-01-06 (Estimated); Last update posted 2016-01-06 (Estimated); Status verified 2016-01

CONDITIONS: Dyspnea
MeSH Terms: conditions — Dyspnea

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 5 Years
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (2):
- pulmonary hypertension: The two groups were defined by catheterization result. (no intervention)
  Interventions: Other: no intervention
- non-pulmonary hypertension: The two groups were defined by catheterization result. (no intervention)
  Interventions: Other: no intervention

INTERVENTIONS:
Other: no intervention — no intervention

SUMMARY:
This study investigated clinical parameters, laboratory data, imaging studies to evaluate patients with suspected pulmonary hypertension.

DETAILED DESCRIPTION:
Left and right ventricular ejection fraction (LV/RV EF) at rest and immediately after exercise treadmill test (ETT) were measured by nuclear medicine study in consecutively symptomatic patients with suspected pulmonary hypertension, along with other clinical variables were correlated with right heart catheterization parameters.

ELIGIBILITY:
Inclusion Criteria:

* patients suspicious for pulmonary hypertension.

Exclusion Criteria:

* pregnant, lactating, CAD history

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients suspicious for pulmonary hypertension
Sampling Method: Probability Sample
Enrollment: 300 (Estimated)
Dates: Start 2009-07; Primary Completion 2018-12 (Estimated); Study Completion 2018-12 (Estimated)

PRIMARY OUTCOMES:
All-cause mortality | an average of 1 year

CONTACTS AND LOCATIONS:
Overall Officials: Mei-Fang Cheng, M.D., Principal Investigator — National Taiwan University Hospital and National Taiwan University College of Medicine
Locations (1):
- National Taiwan University Hospital and National Taiwan University College of Medicine, Taipei, Taiwan